CLINICAL TRIAL: NCT03821454
Title: A Randomized, Double-blind, Placebo-controlled Study of Capecitabine in the Treatment of Early-stage Breast Cancer With Low-hormone Receptor Expression and Residual Invasive Carcinoma After Neoadjuvant Chemotherapy
Brief Title: Capecitabine in the Treatment of Breast Cancer With Low-hormone Receptor Expression After Neoadjuvant Chemotherapy
Acronym: CALORIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CALORIE
Record Dates: First submitted 2019-01-26; First posted 2019-01-29 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine (Experimental): The experimental group received oral capecitabine for eight cycles.
  Interventions: Drug: Capecitabine
- Placebo (Placebo Comparator): The placebo group received oral placebo for eight cycles.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Capecitabine — Oral capecitabine (at a dose of 1250 mg per square meter of body-surface area, twice per day, on days 1 to 14) every 3 weeks for eight cycles.
  Arms: Capecitabine
Drug: Placebos — Oral Placebos (twice per day, on days 1 to 14) every 3 weeks for eight cycles.
  Arms: Placebo

SUMMARY:
Capecitabine is recommended for adjuvant treatment of advanced or metastatic breast cancer and is particularly effective in patients with triple-negative breast cancer (TNBC).

CREATE-X clinical studies have demonstrated that Capecitabine can further improve prognosis and demonstrate good tolerance in patients who have not achieved pathologic complete response (pCR) after neoadjuvant chemotherapy.

Previous studies have confirmed that the pathological features of the low- hormone receptor (HR)positive population in breast cancer are similar to those in the TNBC population, with a poor prognosis and are not sensitive to adjuvant endocrine therapy.

We hypothesize that the use of Capecitabine in breast cancer patients with residual invasive carcinoma after neoadjuvant chemotherapy may improve prognosis.

DETAILED DESCRIPTION:
The investigators will recruit patients who had low- hormone receptor (HR)positive breast cancer of stage I - IIIC and pathologically assessed residual cancer cells (no pathological complete response, non-pCR) after neoadjuvant chemotherapy with anthracycline, taxane, or both. Participants who have residual components of ductal carcinoma in situ are assessed as having a pathological complete response. Participants with tumor-positive lymph nodes excluded.

Other key eligibility criteria are low- hormone receptor (HR)positive, including low-ER and low-PR, low-ER and PR-negative, low-PR and ER-negative. The definition of low hormone receptor (HR) positive is nuclear staining of 1%-10% of the epithelial component of the tumor.

Eligible participants are centrally enrolled after pathological assessment and are randomly assigned in a 1:1 ratio to receive either capecitabine plus standard therapy or standard therapy alone (control).

The trial treatments are standard postsurgical treatments, which included endocrine therapy in participants with estrogen-receptor-positive (nuclear staining ≥ 1%) disease, targeted therapy in participants with HER-2 overexpression and radiotherapy (if indicated), with or without capecitabine.

After surgery, the capecitabine group receive oral capecitabine (at a dose of 1250 mg per square meter of body-surface area, twice per day, on days 1 to 14) every 3 weeks for eight cycles. The concomitant administration of postsurgical endocrine therapy is allowed. Postsurgical radiotherapy could be given before or after randomization and could be concomitant with postsurgical endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Women and men at least 18 years of age or older.
3. Pathological confirmation of breast cancer
4. Tumor stage(TNM): T1-4N0-3M0
5. No evidence of distant metastasis
6. Adequate bone marrow, hepatic, and renal function
7. Measurable disease as per RECIST criteria
8. Karnofsky≥70
9. Laboratory criteria:

PLT≥100*109/L WBC≥4000/mm3 HGB≥10g/dl ALT and AST<2*ULN

Exclusion Criteria:

1. Presence of metastatic disease.
2. Inflammatory breast cancer.
3. Bilateral breast cancer.
4. Postoperative treatment with other adjuvant chemotherapy drugs.
5. Other malignant tumors (concurrent or previous).
6. Pregnant woman.
7. Hypersensitive to any drug in Capecitabine or any ingredient of Capecitabine.
8. Any severe systemic disease contraindicating chemotherapy.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival(DFS) | Time of Surgery up to 5 years.
  First Dose of Capecitabine or Placebo to first documentation of local or distant recurrence, or death or initiation of antineoplastic therapy before documentation of first relapse.
Overall Survival(OS) | First Dose of Capecitabine or Placebo up to 5 years.
  Time from the first dose of Capecitabine or Placebo to death due to any cause.

IPD SHARING:
Plan to Share IPD: No